CLINICAL TRIAL: NCT01930227
Title: Effect of Transcutaneous Electrical Acupoint Stimulation(TEAS) on the Incidence of Hypotension After Spinal Anesthesia in Patients Undergoing Cesarean Section: a Prospective, Randomized Controlled Trial
Brief Title: Transcutaneous Electrical Acupoint Stimulation(TEAS) for Hypotension After Spinal Anesthesia in Parturients
Acronym: THSAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: wangqiang (Other)
Responsible Party: Sponsor-Investigator, wangqiang, Professor, Xijing Hospital
Organization: Xijing Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: XJH-A-2013-08-1
Record Dates: First submitted 2013-08-24; First posted 2013-08-28 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Hypotension
Keywords: hypotension; spinal anesthesia; cesarean
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- TEAS Treatment (Experimental): Patients were given 30min of TEAS at PC6 after spinal anesthesia
  Interventions: Other: TEAS
- Non-acupoint stimulation (Sham Comparator): Patients were given 30min of electrical stimulation at shoulder after spinal anesthesia
  Interventions: Other: Non-acupoint stimulation
- Control (No Intervention): No stimulation was given

INTERVENTIONS:
Other: TEAS — Electric stimulation was given through electrode attached to specific acupoints
  Other Names: Transcutaneous electrical acupoint stimulation
  Arms: TEAS Treatment
Other: Non-acupoint stimulation — Electric stimulation was given through electrode attached to the shoulder
  Arms: Non-acupoint stimulation

SUMMARY:
The purpose of this study is to compare the effect of TEAS on hypotension after spinal anesthesia in patients undergoing cesarean section

DETAILED DESCRIPTION:
Patients were randomly assigned to 3 groups, receiving TEAS , non-acupoint stimulation or no-stimulation after spinal anesthesia respectively. 1.4 ml of bupivacaine mixed with 0.2ml of 50% glucose was given for spinal anesthesia under lateral position. Then the patient was switched to supine position and the OR table was tilted to the left for 15 degree. The sensory loss level was assessed. The blood pressure and heart rate every 2min were recorded for 30min after spinal anesthesia. The adverse events and use of ephedrine adverse events were recorded as well.

ELIGIBILITY:
Inclusion Criteria:

* Age>18yrs
* American Society of Anesthesiologists(ASA) status 1-2
* Scheduled for elective cesarean under spinal anesthesia
* Gestational age>38weeks, singleton pregnancy
* Informed consented

Exclusion Criteria:

* Patients with pre-eclampsia or diabetes
* Patients with hypertension or cardiac dysfunction
* Disturbance of communication
* Placental abruption

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2013-09; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Incidence of hypotension | During 30min after spinal anesthesia

SECONDARY OUTCOMES:
Average systemic blood pressure(SBP) and diastolic blood pressure(DBP) | During 30min after spinal anesthesia
Lowest SBP and DBP | During 30min after spinal anesthesia
Dosage of ephedrine | During 30min after spinal anesthesia
postoperative nausea and vomiting(PONV) score | During 30min after spinal anesthesia
Incidence of dizzy and dyspnea | During 30min after spinal anesthesia
Change of concentration of serum adrenaline and noradrenaline | Immediately after TEAS

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong LU, MD, Principal Investigator — Air Force Military Medical University, China
Locations (2):
- China (2):
  - Women and Children's Hospital of Shaanxi Province, Xi'an, Shaanxi
  - Xijing Hospital, Fourth Military Medical University, Xi'an, Shaanxi

REFERENCES:
- [Background] Sahmeddini MA, Eghbal MH, Khosravi MB, Ghaffaripour S, Janatmakan F, Shokrizade S. Electro-acupuncture stimulation at acupoints reduced the severity of hypotension during anesthesia in patients undergoing liver transplantation. J Acupunct Meridian Stud. 2012 Feb;5(1):11-4. doi: 10.1016/j.jams.2011.11.001. Epub 2011 Dec 7. PMID 22309902
- [Background] Arai YC, Kato N, Matsura M, Ito H, Kandatsu N, Kurokawa S, Mizutani M, Shibata Y, Komatsu T. Transcutaneous electrical nerve stimulation at the PC-5 and PC-6 acupoints reduced the severity of hypotension after spinal anaesthesia in patients undergoing Caesarean section. Br J Anaesth. 2008 Jan;100(1):78-81. doi: 10.1093/bja/aem306. Epub 2007 Oct 24. PMID 17959591
- [Background] Syuu Y, Matsubara H, Hosogi S, Suga H. Pressor effect of electroacupuncture on hemorrhagic hypotension. Am J Physiol Regul Integr Comp Physiol. 2003 Dec;285(6):R1446-52. doi: 10.1152/ajpregu.00243.2003. Epub 2003 Jul 31. PMID 12893654